CLINICAL TRIAL: NCT02621216
Title: Tilburg Health Outcomes Registry of Emotional Stress in Coronary Intervention
Acronym: THORESCI
Status: Recruiting | Type: Observational
Sponsor: Tilburg University (Other)
Collaborators: The Elisabeth-TweeSteden Hospital (Other); Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: Principal Investigator, Nina Kupper PhD, Associate Professor of Medical Psychology, Tilburg University
Other Study IDs: THORESCI; NL46259.028.13 (Other: CCMO)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Coronary Heart Disease
Keywords: percutaneous coronary intervention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background of the study:

Percutaneous coronary interventions (PCI) have become mainstay treatment for acute coronary artery disease and the number of patients receiving PCI is vastly growing. However, relatively little long-term follow-up studies of large real-world clinical samples exist that have looked at the real-world effects of PCI treatment and adherence to current guidelines.

Psychological risk factors are important in determining prognosis after PCI, and undergoing PCI may increase the risk of low mood. To date, studies have examined single psychological risk factors, without taking into account their relatedness. Moreover, guidelines are advocating psychosocial screening in early cardiovascular disease, but the screening test as proposed in the prevention guideline has not yet been validated or tested. Although the detrimental effects of psychological risk factors on cardiovascular prognosis are known, the mechanisms through which they exert these effects are yet unclear. It is to be expected that not one but multiple biological (inflammation, endothelial dysfunction) and behavioural (coping styles, poor self-care, consultation behaviour) pathophysiological processes play a role, and that these processes interact with each other. In PCI patients the mechanisms linking psychological risk to poor prognosis are still to be investigated.

Objective of the study:

1. To examine the adherence to the prevention and PCI guidelines and the effects thereof on long term prognosis in PCI patients.
2. To evaluate the effectiveness of the psychosocial screening instrument of the European Society of Cardiology Prevention guideline 2012.
3. To examine effects of clustering psychological risk factors on several networks of potentially mediating mechanisms and long term outcomes in a large sample of PCI patients.

DETAILED DESCRIPTION:
Rationale: Percutaneous coronary interventions (PCI) have become mainstay treatment for acute coronary artery disease and the number of patients receiving PCI is vastly growing. Clinical trials have reported on the efficacy and effects on quality of life and mortality. Guidelines have been constructed for PCI treatment as well as cardiovascular prevention. However, relatively little long-term follow-up studies of large real-world clinical samples exist that have looked at the real-world effects of PCI treatment and adherence to current guidelines.

Moreover, psychological risk factors are important in determining prognosis after PCI, and undergoing PCI may increase the risk of low mood. To date, studies have examined single psychological risk factors, without taking into account their relatedness. Moreover, guidelines are advocating psychosocial screening in early cardiovascular disease, but the screening test as proposed in the ESC Prevention guideline has not yet been validated or tested.

Although the detrimental effects of psychological risk factors on cardiovascular prognosis are known, the mechanisms through which they exert these effects are yet unclear. It is to be expected that not one but multiple biological (inflammation, endothelial dysfunction) and behavioural (coping styles, poor self-care, consultation behaviour) pathological processes play a role, and that these processes interact with each other. In PCI patients, the mechanisms linking psychological risk to poor prognosis are still to be investigated. Objective: (1) To examine the adherence to the prevention and PCI guidelines and the effects thereof on long term prognosis in PCI patients. (2) To examine effects of clustering psychological risk factors on several networks of potentially mediating mechanisms and long term outcomes in a large sample of PCI patients. (3) To evaluate the effectiveness of the psychosocial screening instrument of the European Society of Cardiology Prevention guideline 2012. Study design: Prospective observational cohort study. Study population: All patients aged >18 admitted to the TweeSteden hospital for percutaneous coronary intervention are eligible. Main study parameters/endpoints: Predictors: Psychological (risk) factors (depression, anxiety, Type D personality, mindfulness, positive mood), Adherence; Outcome variables: PCI complications, hospitalizations, events. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk associated with the current study is very low. For this mechanistic observational study, investigators will ask patients to fill out two extensive (20 pages) and then several smaller (12-15 pages) psychological surveys including among others questions on personality, positive and negative mood, mindfulness, work stress, and satisfaction with life. Preferably, questionnaires will be administered digitally by email link. There are no direct benefits of participation, other than providing data to create knowledge to improve future treatment.

ELIGIBILITY:
Inclusion Criteria:

* PCI
* Sufficient understanding of Dutch language

Exclusion Criteria:

* life threatening comorbidity (e.g., metastasized cancer)
* cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for either elective or (sub-)acute PCI for ≥1 coronary occlusions
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-12-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
PCI complications | 1 year
  procedure related complications, events and mortality in the first year post-PCI

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kupper, PhD, Principal Investigator — Tilburg University
Locations (1):
- Elisabeth-TweeSteden hospital, Tilburg, North Brabant, Netherlands

REFERENCES:
- [Derived] Douma ER, Kop WJ, Kupper N. Associations Between Psychological Factors and Adherence to Health Behaviors After Percutaneous Coronary Intervention: The Role of Cardiac Rehabilitation. Ann Behav Med. 2024 Apr 11;58(5):328-340. doi: 10.1093/abm/kaae008. PMID 38431284

DOCUMENTS (2):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT02621216/Prot_004.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT02621216/SAP_002.pdf